CLINICAL TRIAL: NCT03070574
Title: Mesalamine for Colorectal Cancer Prevention Program in Lynch Syndrome - MesaCAPP
Brief Title: Mesalamine for Colorectal Cancer Prevention Program in Lynch Syndrome
Acronym: MesaCAPP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor patient recruitment and insufficient financing.
Sponsor: Christoph Gasche (Other)
Collaborators: Prof. Dr. Gabriela Möslein, Germany (Unknown); Prof. Dr. Hans Vasen, The Netherlands (Unknown); Prof. Dr. med. Jan Lubinski, Poland (Unknown); Prof. Dr. med. Yaron Niv, Israel (Unknown); Univ. Prof. Dr. Judith Karner-Hanusch, Austria (Unknown); Ann-Sofie Backman, MD PhD, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Christoph Gasche, Univ. Prof. Dr. Christoph Gasche - Coordinating Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MesaCAPP; NCT02864979 (obsolete NCT alias)
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: Lynch Syndrome; Chemoprevention; Mesalazine; 5-ASA
MeSH Terms: conditions — Colorectal Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2400 MG mesalamine (5-ASA) total (Experimental): 2400mg (1200mg mesalamine/1200mg) mesalamine once daily in the morning for the treatment phase of the study (24 months)
  Interventions: Drug: mesalamine 2400 MG (5-ASA)
- 1200 MG mesalamine (5-ASA) total (Experimental): placebo/1200mg mesalamine once daily in the morning for the treatment phase of the study (24 months)
  Interventions: Drug: mesalamine 1200 MG; Other: Placebo
- Placebo (Placebo Comparator): placebo/placebo once daily in the morning for the treatment phase of the study (24 months)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: mesalamine 2400 MG (5-ASA) — For this study IMP will be supplied as film-coated tablets packed in containers. Each patient will receive two different containers, each 1200mg of IMP (= 2400 mg), every 3 months (± 1 week), 100 tablets per container. The containers will be marked in different colours, to prevent the patients from taking two tablets from one container accidentally.
  Other Names: Mezavant; Mesalazine; 5-aminosalicylic acid (5-ASA)
  Arms: 2400 MG mesalamine (5-ASA) total
Drug: mesalamine 1200 MG — For this study IMP will be supplied as film-coated tablets packed in containers. Each patient will receive two different containers of IMP (1200 mg/placebo) every 3 months (± 1 week), 100 tablets per container. The containers will be marked in different colours, to prevent the patients from taking two tablets from one container accidentally.
  Other Names: Mezavant; Mesalazine; 5-aminosalicylic acid (5-ASA)
  Arms: 1200 MG mesalamine (5-ASA) total
Other: Placebo — For this study IMP will be supplied as film-coated tablets packed in containers. Each patient will receive two different containers of IMP (placebo/placebo) every 3 months (± 1 week), 100 tablets per container. The containers will be marked in different colours, to prevent the patients from taking two tablets from one container accidentally.
  Arms: 1200 MG mesalamine (5-ASA) total; Placebo

SUMMARY:
Multicenter, multinational, randomized, 3-arm, double-blind, phase II clinical study with 2400mg mesalamine, 1200mg mesalamine or placebo for prevention of colorectal neoplasia in Lynch Syndrome patients for 2 years.

DETAILED DESCRIPTION:
This is a multicenter, multinational, randomized, 3-arm, double-blind, phase II clinical study with 2400mg mesalamine (5-ASA), 1200mg mesalamine (5-ASA) or placebo in LS patients for a 2-year treatment. 540 tumor free carriers of a known genetic mutation in a major MMR gene (including patients in which the polyps are endoscopically removed) will be randomized 1:1:1 (180 each) to receive 2400mg mesalamine, 1200mg mesalamine or placebo. Patients will be identified through local or national registries and through collaboration with sites. Tumor free patients, assessed by white light high resolution colonoscopy, will be randomized to the study. A serum and stool sample will be taken to identify for mesalamine compliance and potential biomarkers. Biopsies of the normal tissue of ascending colon and rectum will be taken at the first and the last colonoscopy.

The aim of the study is to investigate the effect of regular treatment with mesalamine (5-ASA) on the occurrence of any colorectal neoplasia, tumor multiplicity (the number of detected adenomas/carcinomas) and tumor progression in LS patients.

A 50% reduction of the occurrence of colorectal neoplasia in mesalamine-treated patients is expected. Tumor multiplicity and tumor progression (severity of the neoplastic lesions) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Proven tumor-free (including patients in which the polyps are removed endoscopically) carriers of a germline pathologic mutation on one of the MMR genes including MLH1, MSH2 (including EpCAM) and MSH6
* Male or female subjects with the age > 25 years
* Females who have been post-menopausal more than one (1) year or females of childbearing potential using a highly efficient method of contraception with less than 1% failure rate (i.e. oral hormonal contraceptives, hormone implants, hormone injections, sterilization, hormonal or copper intrauterine device, sterilized/vasectomized partner, or diaphragm in combination with a condom, spermicide or birth control pills) or should agree to abstain from heterosexual activity during treatment period. Females of childbearing potential must have a negative pregnancy test at screening and before randomization.
* Signed written informed consent prior to inclusion in the study

Exclusion Criteria:

* Presence of colorectal endoscopically non-removable benign neoplasia (patient can be included if the adenoma is removed)
* Carriers of germline mutations in PMS2
* Patients with history of stage 3 and 4 colorectal cancer (CRC) are excluded
* Presence of metastatic disease
* Regular use of acetylsalicylic acid (ASA or aspirin): daily use of ≥100mg in more than 3 continuous months within the last year
* Regular use of NSAIDs or COX-2 inhibitors: daily use in more than 3 continuous months within the last year
* Hypersensitivity to 5-ASA
* Patients after total or subtotal colectomy
* Colorectal surgery within the previous 6 months
* Unwillingness to participate or who is considered incompetent to give an informed consent
* Pregnant or breastfeeding women
* Participation in another clinical study investigating another IMP within 3 months prior to screening
* Renal insufficiency (GFR <30ml/min/1.73m2)
* Severe liver disease or liver failure (elevation of liver enzymes above 3xULN)
* Current or history of serious psychiatric disorder or alcohol/drug abuse that in the opinion of the investigator may impact the assessment of IMP safety andefficacy or protocol adherence
* Prior history of myocarditis or pericarditis. Other severe acute or chronic medical condition (such as severe chronic lung (COPD, including asthma), kidney or heart diseases) or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or ability to comply with study procedures, IMP administration and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Reduction in the occurrence of any colorectal neoplasia in LS patients | End of treatment at 24 months +/- 1 month
  • Occurrence of any colorectal neoplasia (both benign and malignant tumors) between groups is described by absolute frequencies and percentages with 95 % confidence intervals. A logistic regression is used to assess differences between active treatment and placebo for the occurrence of any colorectal neoplasia, adjusted for country and history of cancer before randomization. Treatment effects are assessed by odds-ratios and corresponding 95 % confidence intervals.
Reduction in the occurrence of any colorectal neoplasia in LS patients | End of study at year 6 +/- 3 months
  As above

SECONDARY OUTCOMES:
Tumor multiplicity | End of treatment at 24 months +/- 1 month
  The number of colorectal neoplasia (both benign and malignant tumors) per patient will be tested between groups by an analysis of variance, adjusting for country and history of cancer before randomization. In case of non-normally distributed residuals a suitable transformation to achieve normal distribution is considered.
  It will be tested whether 5-ASA (low- and high-dose together) reduces the number of any colorectal neoplasia (both benign and malignant tumors; tumor multiplicity) compared to placebo in LS patients at the end of treatment and end of study. Advanced adenomas are defined by a diameter above 1 cm villous or tubulo-villous histology or high grade dysplasia.
  All tests are two-sided and a significance level of 5 % is used.
Tumor progress | End of treatment at 24 months +/- 1 month
  The tumor progress in 4 ordered stages will be tested between groups by a chi-square trend test stratified for country and history of cancer before randomization and modelled by an ordinal logistic regression.
  It will be tested whether 5-ASA (low- and high-dose together) reduces tumor progression (compared 4 ordinal stages: no colorectal neoplasia / non-advanced adenoma / advanced adenoma / carcinoma) compared to placebo in LS patients at the end of treatment and end of study. Advanced adenomas are defined by a diameter above 1 cm villous or tubulo-villous histology or high grade dysplasia.
  All tests are two-sided and a significance level of 5 % is used.
Treatment effects | End of treatment at 24 months +/- 1 month
  The dependence of treatment effects on history of colorectal cancer, sex and patients age (<45 years and ≥45 years) will be assessed by modelling interactions between these factors and treatment in the corresponding regression models.
  If differences between 5-ASA (low- and high-dose together) effects and placebo effects on the occurrence of colorectal neoplasia, tumor multiplicity or tumor progression depend on the history of colorectal cancer, sex and patients age (LS patients below 45 years of age or 45 years of age and older) will be investigated.
  All tests are two-sided and a significance level of 5 % is used.
High and low dose ASA | End of treatment at 24 months +/- 1 month
  Differences between high and low dose ASA for the occurrence of colorectal neoplasia, tumor multiplicity and tumor progression will be analysed by the same methods as for the comparison between ASA and placebo to investigate differences between low and high dose 5-ASA with respect to the occurrence of colorectal neoplasia, to tumor multiplicity and tumor progression.
  All tests are two-sided and a significance level of 5 % is used.
Significant findings & illnesses - adverse events | End of treatment at 24 months +/- 1 month
  Safety data are described and compared between groups in an exploratory manner to determine the safety concerning 5-ASA in LS patient. Therefore significant findings/illnesses, reported after the start of the study and which meet the definition of an AE, will be recorded in the CRF.
  Intention to treat set: This analysis set includes subjects who were randomized (and received at least one dose study drug). This analysis set will be chosen for safety assessment.
  All tests are two-sided and a significance level of 5 % is used.

CONTACTS AND LOCATIONS:
Locations (6):
- Department of Surgery, Medical University Vienna, Vienna, Austria
- HELIOS Universitätsklinikum Wuppertal, Zentrum für Hereditäre Tumorerkrankungen, Wuppertal, North Rhine-Westphalia, Germany
- Rabin Medical Center Beilinson Hospital Gastroenterology Department, Petah Tikva, Israel
- Leiden University Medical Center, Leiden, Netherlands
- Department of Genetics and Pathomorphology of Pomeranian Medical University, Szczecin, Poland
- Karolinska universitetsjukhuset, A6:00 Gastroenterologiskt öppenvårdscentrum, Mottagningen för ärftlig tarmcancer, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No